CLINICAL TRIAL: NCT01842698
Title: Feasibility of the Use of Ultrasound-guided Paravertebral Catheterisation for the Analgesic Management of Thoracotomy
Brief Title: Ultrasound-guided PVB
Acronym: BPV échoguidé
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped because there was a technical problem with the ultrasound used in the trial.
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPVéchoguidé
Record Dates: First submitted 2013-02-14; First posted 2013-04-30 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Thoracotomy Surgery; Anesthesia; Ultrasound-guided PVB; Post-operative Pain
Keywords: Thoracotomy surgery; Anesthesia; Ultrasound-guided PVB; Post-operative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ultrasoundguided paravertebral catheter (Experimental): ultrasoundguided paravertebral catheter
  Interventions: Device: ultrasoundguided paravertebral catheter

INTERVENTIONS:
Device: ultrasoundguided paravertebral catheter
  Other Names: ultrasound-guided paravertebral catheterisation

SUMMARY:
Thoracotomy, is a surgical procedure performed routinely in connection with pulmonary surgery. Pain induced by thoracotomy is considered as the most severe post-operative pain. Control of the pain is essential in the perioperative management.

Nowadays, there are several strategies to support this pain, including regional anesthesia techniques in the context of multimodal analgesia. Epidural analgesia reduces pain scores and respiratory complications significantly. ParaVertebral Block (PVB) is a technique as effective as epidural analgesia in the treatment of pain after thoracotomy and could present a more limited number of complications. However, there is no consensus on the best technique for realisation of PVB.

Para-vertebral catheterisation can be performed by posterior approach in seeking a strength loss after bone contact of transverse vertebral process using the technique of Eason and Wyatt, but it is a blind technique. The ultrasonographic control, developed in the context of all puncture invasive actions, is an effective contribution to the realisation of a BPV, but still insufficiently validated. First used to measure the distance skin - posterior costo-transverse ligament and skin - parietal pleura before procedure, the ultrasonography has recently led to the publication of echo-guided techniques combining recognition of structures defining the space para- vertebral, viewing the progression of the needle and the spread of the local anesthetic. The handling of the ultrasonographic probe associated with the puncture requires additional learning.

The objective of this project is to study the feasibility of para-vertebral catheter insertion under ultrasonographic control. The appearance like "pigtail" of the catheter, the most recently proposed, seems the more attractive in terms of safety. The aim of this pilot prospective study is accurately quantify all qualitative parameters related to the technique in order to achieve a future validation with a medico-economic component.

Ultrasound-guided technique will correspond to a technique with a puncture of the lateral to medial space described by Shibata, after spotting of the first rib proposed by Bouzinac.

This study will be proposed to patients undergoing thoracotomy for total or partial pulmonary resection in Thoracic Surgery service of Centre Jean Perrin, the number of patients required is 60 patients over a period of inclusion of 12 months.

DETAILED DESCRIPTION:
Prospective followed of cohort including consecutive patients, all receiving the same technique of anesthesia and analgesia:

* Preoperative para-vertebral catheterisation on the surgery side.
* Preoperative test of the efficiency of para-vertebral block.
* Conventional general anesthesia.
* Conventional rescue postoperative analgesia.
* Systematic radiographic control with injection of contrast product into the para-vertebral catheter.
* Conventional postoperative monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing programmed lateral or posterolateral thoracotomy, regardless of indication,
* Aged 18 to 80 years

Exclusion Criteria:

* Surgery performed in the emergency;
* Specific clinical contexts including neoplasia in terminal phase or palliative phase;
* Contraindications to the products of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The overall failure rate of the para-vertebral block | 24 hours
  The overall failure rate of the para-vertebral block ( failed installation or efficiency)

SECONDARY OUTCOMES:
The time (in minutes) between the start of the installation and the effective para-vertebral block obtaining | 24 hours
  Effective para-vertebral block obtaining
Paravertebral block catheterisation | 24 hours
  •Paravertebral catheterisation efficiency
Paravertebral block efficiency | 24 hours
  Paravertebral block efficiency
Pain evaluation | H0+30 min, +1h, +1h30, +2h, +4h, +8h, +12h, +16h, +20h, +24h, +32h, +40h, +48h
  •Pain evaluation with Analogic Visual Scale
Tolerance hemodynamic, nausea and vomiting | 72 hours
  Tolerance hemodynamic, nausea and vomiting reporting

CONTACTS AND LOCATIONS:
Overall Officials: Hammou TAHERI, PhD, Principal Investigator — Centre de lutte contre le cancer - Centre Jean Perrin
Locations (1):
- Centre de lautte contre le cancer - Centre Jean Perrin, Clermont-Ferrand, France